CLINICAL TRIAL: NCT03447015
Title: Effects of Ambulation During First Stage of Labour on Maternal and Neonatal Outcomes: A Randomized Controlled Trial
Brief Title: Effects of Ambulation During First Stage of Labour on Maternal and Neonatal Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Reham Mohammad Khresheh, Dr. Reham Khresheh, Mutah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 112018
Record Dates: First submitted 2018-02-12; First posted 2018-02-27 (Actual); Results first posted 2019-10-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2019-09

CONDITIONS: Labor Pain
Keywords: ambulation; labour; Randomized Controlled Trial; Jordan
MeSH Terms: conditions — Labor Pain | interventions — Walking

STUDY DESIGN:
Intervention Model Description: A randomised controlled study will be conducted with primiparous women. In the intervention group women will be encouraged to ambulate and women in the control group will receive usual maternity care
Who Masked: Investigator
Masking Description: The principal researcher will be kept blind for those participants who are in the intervention and control groups. Completing the second part of the study tool, which is related to maternal and infant health outcomes, will be in maternal ward and by the primary investigators 24 to 48 hours after birth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulation during labour (Experimental): women will be encouraged to ambulate "Ambulation during labour" here will refer to moving from place to place during the first stage of labour that reduces the amount of time a woman spends laying down during this stage (measured by recording the number of minutes spend on walking).
  Interventions: Other: ambulation
- Standard Maternity care (No Intervention): women will receive usual maternity care.

INTERVENTIONS:
Other: ambulation — "Ambulation during labour" here will refer to moving from place to place during the first stage of labour that reduces the amount of time a woman spends laying down during this stage (measured by recording the number of minutes spend on walking).
  Arms: Ambulation during labour

SUMMARY:
This study investigates the effect of ambulation (walking) during first stage of labour on maternal and neonatal outcomes. In the intervention group women will be encouraged to ambulate and women in the control group will receive usual maternity care.

DETAILED DESCRIPTION:
Walking and upright positions in the first stage of labour reduces the duration of labour, the risk of caesarean birth, and the need for epidurals. Movement is a safe and healthy coping strategy for pain, and confining labouring women to bed increases pain and decreases women's satisfaction with their birth experience . Despite that ambulation and upright positioning during labour does not harm mother, fetus, or newborn, women are still largely confined to bed during the first stage of labour. The increased use of medical interventions such as epidural analgesia, continuous electronic fetal monitoring, intravenous infusions for fluids and electrolytes, and a restrictive birthing environment limits women's instinctive responses to labour pain and contractions rather than assisting the woman to cope with the pain and anxiety of labour .

In Jordan practices in maternity wards are not based on best evidence.The majority of health facilities restrict movement during labour, women were confined to bed in the lithotomy position and most of these facilities strap women in the delivery position, women have no choice to assume the position they prefer during labour and delivery. The practice of restricting women's movement in labour is contrary to the statements and recommendations of professional organizations advocate for women to move about during the first stage of labour, as long as they remain low-risk. Implementing evidence-based maternity care in developing countries with limited resources such as Jordan is particularly challenging, and requires commitment to applying the most up to date evidence to clinical decisions.

The purpose of this study is to begin investigation that could help provide a better quality of care during birth and improve maternity outcomes in one Jordanian hospital. The process was introducing an evidence-based practice of encouraging women to ambulate and assume the upright position during the first stage of labour and observing if results would suggest low cost modifications for the maternity health service environment, especially the labour ward. This is the first study that has attempted to implement and evaluate such an intervention in Jordan.

Methods A randomised controlled study will be conducted with primiparous women who come to give birth at Al- Karak Hospital in Jordan. Women will be subsequently randomised into the groups using a table of random numbers. "Ambulation during labour" here will refer to moving from place to place during the first stage of labour that reduces the amount of time a woman spends laying down during this stage (measured by recording the number of minutes spend on walking).

The setting for this study will be the maternity ward at Al-Karak hospital, the main governmental and teaching hospital in the southern region of Jordan. In 2016 2,808 births occurred in this hospital, 59% were caesarean births . In this hospital, the woman usually labours in 26- bed ward with restrictions on movement. This is consistent practice nationally. Certified midwives, resident physicians, and obstetricians provide care. Midwives in this hospital work with uncomplicated labours and help obstetricians with complicated cases.

The sample size was calculated using the G power version 3.1. Based on difference between two independent groups, alpha= 0.05, median effect size 0.3, power =95%, sample size required for each group is 88 women. To overcome attrition, 25% of the calculated sample will be added, the final sample size will be 110 women in each group.

Data will be collected using structured tool developed by the researchers based on literature review of research related to the current topic. The tool composed of section collecting the socio-demographic data and another section collecting maternal and neonatal outcomes. The research tool was reviewed by a panel (n=3) of experts in maternity health field. Before starting the study, the final version of the tool will be tested in a pilot study to evaluate its feasibility, clarity, and reliability. Assistant researcher (midwife) will complete the first section of the tool, which related to socio-demographic data, and will allocate participants to control and intervention group according to the randomization list. The principal researcher will be kept blind for those participants who are in the intervention and control groups. Completing the second part of the study tool, which is related to maternal and infant health outcomes, will be in maternal ward and by the primary investigators 24 to 48 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women
* with uncomplicated singleton pregnancies
* between 37 and 41 weeks gestation, cephalic, with cervical dilatation 3 to 5cm

Exclusion Criteria:

* multiparous
* with complicated pregnancies , multiple gestation,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All primiparous women with uncomplicated singleton pregnancies between 37 and 41 weeks gestation, cephalic, with cervical dilatation 3 to 5cm who come to give birth at Al-Karak hospital, between the 1st of January and the 30th of December 2018 will be approached for participation
Enrollment: 290 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Khresheh, PhD, Principal Investigator — Mutah University
Locations (1):
- Ministry Of Health, Karak, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bala, I., M. Babu, et al. Effectiveness of Back Massage versus Ambulation During First Stage of Labour among Primigravida Mothers in Terms of Pain and Anxiety. International Journal of Nursing Education 9(3): 28-32, 2017
- [Background] Khresheh R, Homer C, Barclay L. A comparison of labour and birth outcomes in Jordan with WHO guidelines: a descriptive study using a new birth record. Midwifery. 2009 Dec;25(6):e11-8. doi: 10.1016/j.midw.2007.10.007. Epub 2007 Dec 26. PMID 18155816
- [Background] Lawrence A, Lewis L, Hofmeyr GJ, Styles C. Maternal positions and mobility during first stage labour. Cochrane Database Syst Rev. 2013 Oct 9;2013(10):CD003934. doi: 10.1002/14651858.CD003934.pub4. PMID 24105444
- [Background] Ministry of Health. Health Indicators.http://www.moh.gov.jo/reports. Retrieved 30 September, 2017.
- [Background] Miquelutti, M. A., J. G. Cecatti, et al. The vertical position during labor: pain and satisfaction. Revista Brasileira de Saúde Materno Infantil 9 (4): 393-398, 2009
- [Background] Ondeck M. Healthy birth practice #2: walk, move around, and change positions throughout labor. J Perinat Educ. 2014 Fall;23(4):188-93. doi: 10.1891/1058-1243.23.4.188. PMID 25411538
- [Background] Prabhakar, D., L. S. George, et al. Effectiveness of Ambulation during First Stage of Labour, on the Outcome of Labour among Primigravid Women in Selected Hospitals of Palakkad District, Kerala. International Journal of Nursing Education 7(1): 1-6,2015
- [Background] Romano AM, Lothian JA. Promoting, protecting, and supporting normal birth: a look at the evidence. J Obstet Gynecol Neonatal Nurs. 2008 Jan-Feb;37(1):94-104; quiz 104-5. doi: 10.1111/j.1552-6909.2007.00210.x. PMID 18226163
- [Background] Savitha, V., S. Nayak, et al. Effect of Ambulation during First Stage of Labor on Labor Pain and Outcome of Labor among the Primigravida Mothers in a Selected Hospital Mangalore. Journal of South Asian Federation of Obstetrics and Gyneacology 5(1): 1-3, 2013
- [Background] Shaban IA, Hatamleh R, Khresheh R, Homer C. Childbirth practices in Jordanian public hospitals: consistency with evidence-based maternity care? Int J Evid Based Healthc. 2011 Mar;9(1):25-31. doi: 10.1111/j.1744-1609.2010.00197.x. PMID 21332660
- [Background] Simkin P, Bolding A. Update on nonpharmacologic approaches to relieve labor pain and prevent suffering. J Midwifery Womens Health. 2004 Nov-Dec;49(6):489-504. doi: 10.1016/j.jmwh.2004.07.007. PMID 15544978
- [Background] Souza JP, Miquelutti MA, Cecatti JG, Makuch MY. Maternal position during the first stage of labor: a systematic review. Reprod Health. 2006 Nov 30;3:10. doi: 10.1186/1742-4755-3-10. PMID 17137501
- [Background] Sweidan M, Mahfoud Z, DeJong J. Hospital policies and practices concerning normal childbirth in Jordan. Stud Fam Plann. 2008 Mar;39(1):59-68. doi: 10.1111/j.1728-4465.2008.00151.x. PMID 18540524
- [Background] WHO. Care in normal birth: Apractical guide,1996 .http://www.who.int/maternal_child_adolescent/documents/who_frh_msm_9624/en/.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: women will be encouraged to ambulate "Ambulation during labour" here will refer to moving from place to place during the first stage of labour that reduces the amount of time a woman spends laying down during this stage (measured by recording the number of minutes spend on walking).
  ambulation: "Ambulation during labour" here will refer to moving from place to place during the first stage of labour that reduces the amount of time a woman spends laying down during this stage (measured by recording the number of minutes spend on walking).
- Control: women will receive usual maternity care.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 140 | 150
Completed | 95 | 106
Not Completed | 45 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 95 | 106 | 201
Age, Customized [Number; unit: participants]
  <20 | 10 | 19 | 29
  20-29 | 66 | 79 | 145
  30-39 | 19 | 8 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 106 | 201
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants]
  illiterate | 1 | 21 | 22
  primary school | 11 | 19 | 30
  secondary school | 23 | 22 | 45
  Diploma | 16 | 22 | 38
  Bachelor | 44 | 22 | 66
Employment [Count of Participants; unit: Participants]
  employed | 25 | 17 | 42
  not employed | 70 | 89 | 159
Nationality [Count of Participants; unit: Participants]
  Jordanian | 85 | 106 | 191
  non Jordanian | 10 | 0 | 10
monthly Income (Jordanian Dinar) [Count of Participants; unit: Participants]
  < 200 | 16 | 21 | 37
  200-399 | 11 | 25 | 36
  400-599 | 57 | 55 | 112
  600 and more | 11 | 5 | 16
Residence [Count of Participants; unit: Participants]
  city | 50 | 38 | 88
  village | 45 | 68 | 113
Health insurance [Count of Participants; unit: Participants]
  yes | 54 | 55 | 109
  No | 41 | 51 | 92

OUTCOME MEASURES:

1. Primary Outcome: Duration of the First Stage of Labour
Description: Labour duration will be measured in minutes.
Time Frame: from 3-4 cm of cervical dilatation until delivery of the child.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 106
minutes | 548.337 (62.7841) | 719.585 (86.5829)

2. Primary Outcome: Labour Pain Intensity
Description: Visual Analogue pain Scale rating from 0 to 10 in which the woman registers the pain perception, considering 0 no pain and 10 the worst pain imaginable.)
Time Frame: from time of 4 cm cervical dilatation to to time of full crvical dilatation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 106
Participants
  participants reporting pain intensity as moderate | 26 | 9
  participants reporting pain intensity as severe | 57 | 62
  participants reporting pain intensity very severe | 12 | 35

3. Primary Outcome: Use of Analgesics
Description: used analgesics or did not use
Time Frame: 24 to 48 hours after birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 106
Participants
  yes | 44 | 82
  no | 51 | 24

4. Primary Outcome: Mode of Birth
Description: (defined as normal, vacuum extraction, forceps delivery, or cesarean section)
Time Frame: assessed up to child delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 106
Participants
  number of participants who gave birth normal | 95 | 97
  number of participants who gave birth by vacuum | 0 | 5
  number of participants who gave birth bycesarean | 0 | 4

5. Primary Outcome: Woman's Satisfaction With the Birth Experience
Description: Birth satisfaction scale is a Likert-type scale which is scored according to the responses as indicated: I Strongly Agree. 5; I Agree. 4; I Neither Agree or Disagree: 3; • I Disagree.2; • I Strongly Disagree: 1. The scale consists of 30 items, and total number of scores to be obtained from the scale range between 30, and 150 points. As the scores obtained from the scale increase, level of birth satisfaction increases.
Time Frame: 24 to 48 hours after birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 106
Participants
  Satisfied | 89 | 9
  dissatisfied | 6 | 97

6. Secondary Outcome: Newborn Health Status
Description: measured by Apgar score. Apgar score is a method to quickly summarize the health of newborn. The Apgar scale is determined by evaluating the newborn baby on five simple criteria (Appearance, Pulse, Grimace, Activity, Respiration) on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low
Time Frame: at 5 min of birth of baby
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 106
Participants
  Apgar score ≤ 3 | 2 | 13
  Apgar score 4-6 | 2 | 10
  Apgar score ≥7 | 91 | 83

ADVERSE EVENTS:
Time Frame: 1 year
Description: Any untoward or unfavorable medical occurrence in a participant, considered related to the participant's participation in the research.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/106
Other Adverse Events (participants affected / at risk) | 0/95 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT03447015/Prot_SAP_000.pdf